CLINICAL TRIAL: NCT01687816
Title: Prospective, Nasal Specimen Collection Study in Patients Presenting With Influenza Like Illness and/or Acute Respiratory Infection in an Outpatient Setting
Brief Title: Nasal Specimen Collection Study in Patients With ILI and/or ARI in an Outpatient Setting
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lieselot Houspie (Other)
Responsible Party: Sponsor-Investigator, Lieselot Houspie, PhD student Laboratory of Clinical Virology, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S53729
Record Dates: First submitted 2012-09-06; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Influenza-like Illness; Influenzal Acute Respiratory Infection
Keywords: Influenza-Like-Illness; nasal swabs; Detection of influenza; sensitivity of detection assays

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs of left and right nostril
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No interventions to be administered: Only a nasal swab is collected, no therapeutic interventions

SUMMARY:
This is a prospective specimen collection study targeting patients presenting with Influenza Like Illness (ILI) and/or Acute Respiratory Infection (ARI) in an out-patient setting. A non-invasive, user friendly sampling technique, using midturbinate flocked swabs will be used. These nasal swabs will be collected in different volumes of viral transport media (0.5mL and 3.0mL), for different dilution range of the viruses present in the collected biological specimen. The collection of nasal swabs samples will support the optimization of point of care detection methods for respiratory viruses responsible for ILI and/or ARI.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* All Ages
* Valid Informed Consent and/or Assent, where applicable
* Onset of ILI and/or ARI within the last 3 days (≤ 72h)
* Patient presented with ILI and/or ARI

Exclusion Criteria:

* Invalid Informed Consent and/or Assent
* Onset of ILI and/or ARI was > 3 days (> 72 h)
* Patient did not presented with neither ILI or ARI
* Patient received intranasal attenuated influenza virus in last 3 weeks (example FluMist®, Fluenz®)
* Patient received treatment with influenza direct antivirals in the last 7 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ILI will present with a sudden onset of symptoms and at least one of the following four symptoms: fever or feverishness, malaise, headache, myalgia and at least one of the following three respiratory symptoms: cough, sore throat, shortness of breath.
  Patients with ARI will present with a sudden onset of symptoms and at least one of the following four respiratory symptoms: cough, sore throat, shortness of breath, coryza and the GP's judgment that the illness is due to an infection.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Nasal swab collection of left and right nostril | 1 day
  At the moment volunteer presents him/herself to the general practioner with influenza-like-illness

SECONDARY OUTCOMES:
Completion of questionnaire | 1 day
  Competion of a short questionnaire by the GP recording the clinical symptoms of the patient with ILI

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van Ranst, M.D., PhD, Principal Investigator — Rega Institute, Clinical Virology, Minderbroedersstraat 10, 3000 Leuven
Locations (1):
- University of Leuven (KUL), Leuven, Belgium

REFERENCES:
- [Background] Potter CW. A history of influenza. J Appl Microbiol. 2001 Oct;91(4):572-9. doi: 10.1046/j.1365-2672.2001.01492.x. No abstract available. PMID 11576290